CLINICAL TRIAL: NCT05053308
Title: Proportional Dose of Sublingual Fentanyl Tablet Based on Daily Opioid Requirement Versus Intravenous PCA for Breakthrough Cancer Pain: A Prospective, Randomized, Open Label, Non Inferiority Trial
Brief Title: Proportional Dose of Sublingual Fentanyl Tablet Based on Daily Opioid Requirement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The supply of IP is disrupted
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Associate Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-144-1183
Record Dates: First submitted 2021-08-30; First posted 2021-09-22 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Cancer Pain; Breakthrough Pain
MeSH Terms: conditions — Cancer Pain; Breakthrough Pain | interventions — Infusions, Intravenous; Passive Cutaneous Anaphylaxis; Administration, Sublingual

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV PCA (proportional dosage) (Active Comparator): Breakthrough pain control by bolus based IV patient-controlled anagesia Fentanyl bolus = MME * 15%
  Interventions: Drug: Intravenous Infusion
- SL-FTN (equivalent dose for PCA bolus) (Experimental): Breakthrough pain control by sublingual fentanyl Fentanyl 100mcg/200mcg/300mcg according to the around-the-clock opioid requirement.
  Interventions: Drug: Sublingual Tablet

INTERVENTIONS:
Drug: Intravenous Infusion — IV PCA(fentanyl) Fentanyl bolus = MME * 15%
  Other Names: PCA
  Arms: IV PCA (proportional dosage)
Drug: Sublingual Tablet — subligual fentanyl(Narco®) Fentanyl 100mcg/200mcg/300mcg according to the around-the-clock opioid requirement.
  Other Names: sublingual
  Arms: SL-FTN (equivalent dose for PCA bolus)

SUMMARY:
Proportional dose of sublingual fentanyl tablet (Narco®) based on daily opioid requirement versus intravenous PCA for breakthrough cancer pain: A prospective, randomized, open-label, noninferiority trial.

DETAILED DESCRIPTION:
Based on the previous around-the-clock analgesic demand compared to IV PCA in cancer pain patients to prepare the basis for the administration of fentanyl sublingual tablets with an initial dose.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-80
* Cancer pain
* Admission for the control of cancer pain or consultation for the treatment of cancer pain
* Stable vital sign
* ECOG status ≤ 3 for more than 1 or 2 months
* Opioid-tolerant state
* No history of using sublingual fentanyl

Exclusion Criteria:

* Noncancer pain
* Opioid naive
* baseline NRS pain score> 4
* Current using sublingual fentanyl
* Difficult to assess cancer pain
* no evidence of disease(cancer)
* Planned surgical resection of cancer
* Allergy to fentanyl
* Severe renal and/or liver function
* Severe respiratory depression or uncontrolled COPD

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 11-point scale NRS pain score | 30 minutes after administration
  Change in pain score compared to baseline Score '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"

SECONDARY OUTCOMES:
Change in 11-point scale NRS pain score | 15, 45, 60 minutes after administration
  Change in pain score compared to baseline Score '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"
sum of pain intensity difference(SPID) | 60 minutes after administration
  sum of pain intensity change compared to baseline difference
number of additional doses | immediately after the intervention
  number of additional doses fentanyl bolus or subligual
Pain interference | immediately after the intervention
  Pain interference using BPI-SF
Insomnia | immediately after the intervention
  The severity of insomnia using ISI
Depression | immediately after the intervention
  The severity of depression using Beck Depression Inventory(BDI) 1-10: These ups and downs are considered normal 11-16: Mild mood disturbance 17-20: Borderline clinical depression 21-30: Moderate depression 31-40: Severe depression over 40: Extreme depression
Satisfaction scale | immediately after the intervention
  Satisfaction check using 5 Likert-scale
  (1) Very dissatisfied; (2) Not satisfied; (3) Neutral; (4) Satisfied; (5) Very satidfied

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youn Moon, MD, PhD, Study Chair — Seoul National University Hospital